CLINICAL TRIAL: NCT00422045
Title: Assessment of Low Level Laser Therapy for Late Postoperative Pain After Lumbar Fusion Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xMUO-05
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Surgery
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): No Laser done. All outcome measures are the same.
- 1 (Experimental): Low Level Laser Therapy
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — Low Level Laser Therapy done after surgery.
  Arms: 1

SUMMARY:
The primary objective of this study is to assess whether or not low level laser therapy (LLLT) decreases pain in post-operative orthopedic patients following lumbar fusion surgery.

DETAILED DESCRIPTION:
Lumbar fusion surgery patients typically experience significant post-operative pain for several weeks and their rehabilitation does not start until 8 - 12 weeks postoperatively. We hypothesize that LLLT beginning 4 weeks postoperatively will provide significant reduction in postoperative pain.

ELIGIBILITY:
Inclusion Criteria

* Age > 18 and < 85 years
* Post-operative lumbar fusion surgery
* Currently resides within 100 miles of UMC

Exclusion Criteria

* Pregnant
* Pacemaker
* Medications that have heat or light-sensitivity contraindications (such as: steroids, some antibiotics)
* Two or more cardiac risk factors
* Intraoperative complications
* Wound infection
* Spinal fluid leakage
* Open wound

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
FACES Pain Rating Scale | baseline (2 weeks after surgery), then 6,12, and 24 weeks from baseline
Oswestry Low Back Pain Disability (ODQ) Questionnaire | baseline visit (2 weeks after the patient's surgery date) then 6,12, and 24 weeks thereafter
Quality of Life - The Quality of Life Short-Form Survey (SF-36) | baseline visit (2 weeks after the patient's surgery date) then 6,12, and 24 weeks thereafter

SECONDARY OUTCOMES:
Pain medication usage | baseline (2 weeks after surgery), then 6,12, and 24 weeks from baseline
Improvement measured by serial photographs of surgery appearance and rate of healing | 2 weeks after surgery, then 6, 12, and 24 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Biyani, MD, Principal Investigator — University of Toledo Health Science Campus
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States